CLINICAL TRIAL: NCT05296083
Title: A Safety/Tolerance Phase, Ascending Single Dose Study to Evaluate the Safety and Tolerability of G3P-01, a Food-Grade Pectic Product, in Healthy Volunteers
Acronym: G3P-01-01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SQ Innovation, Inc. (Industry)
Collaborators: EB Medical Research (Unknown); Quartesian (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: G3P-01-01; NL80001.028.21 (Other: CCMO)
Record Dates: First submitted 2022-02-08; First posted 2022-03-25 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Gastrointestinal Discomfort; Performance Status
Keywords: Gastrointestinal; Performance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- G3P-01 50mg Dose Treatment Period 1 (Experimental): G3P-01 will be administered orally as a powdered mixed with water. Treatment Period one dose will be 50mg of IP.
  Interventions: Dietary Supplement: G3P-01
- G3P-01 500mg Dose Treatment Period 2 (Experimental): G3P-01 will be administered orally as a powdered mixed with water. Treatment Period two dose will be 500mg of IP.
  Interventions: Dietary Supplement: G3P-01
- G3P-01 1000mg Dose Treatment Period 3 (Experimental): G3P-01 will be administered orally as a powdered mixed with water. Treatment Period three dose will be 1000mg of IP.
  Interventions: Dietary Supplement: G3P-01
- G3P-01 2000mg Dose Treatment Period 4 (Experimental): G3P-01 will be administered orally as a powdered mixed with water. Treatment Period four dose will be 2000mg of IP.
  Interventions: Dietary Supplement: G3P-01

INTERVENTIONS:
Dietary Supplement: G3P-01 — G3P-01 is a food-grade pectic product derived from squash.

SUMMARY:
This is an interventional, open-label study to evaluate the safety, tolerability and PK of escalating single doses of G3P-01 in 10 healthy adult subjects. All participants will receive G3P-01 in sequential, escalating doses of 50mg (Period 1), 500mg (Period 2), 1,000mg (Period 3), and 2,000mg (Period 4). A wash out period of at least 7 days will occur between doses in each sequential treatment period. Subjects will be admitted Day 1 and stay overnight until the morning of Day 2 for each treatment period. There will be a follow up call 14 days (+/- 2 days) following the last dose of the IP.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged ≥ 18 to < 65 years;
2. Healthy volunteers, as determined by a comprehensive clinical assessment performed at screening (medical history, vital signs, clinical laboratory testing, ECG, and general physical examination);
3. Maintains a regular (mixed or vegetarian/vegan) diet.
4. Non-pregnant, non-lactating females who are either post-menopausal (natural or surgical) or are using at least one (1) of the following forms of contraception:

   * Intrauterine device (IUD),
   * Implantable progestogen-only hormone contraception associated with inhibition of ovulation,
   * Intrauterine hormone-releasing system (IUS),
   * Bilateral tubal occlusion
   * Vasectomized partner
   * Male or female condom with or without spermicide,
   * Cervical cap, diaphragm, or sponge with spermicide,
   * A combination of male condoms with either cervical cap, diaphragm, or sponge with spermicide (double-barrier methods)
   * Combined (estrogen- and progestogen-containing) hormonal contraception associated with inhibition of ovulation

     * oral
     * intravaginal
     * transdermal
     * injectable
   * Progestogen-only hormone contraception associated with inhibition of ovulation

     * oral
     * injectable
   * Abstinence;
5. Willing to adhere to the prohibitions and restrictions specified in the protocol;
6. Must be competent to understand the nature of the study and capable of giving written informed consent and be willing to report for the scheduled study visits and communicate to study personnel about adverse events and concomitant medication use.

Exclusion Criteria:

1. History of any clinically significant cardiac, endocrine, gastrointestinal, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, or renal disease, or other major disease, as determined by the Investigator;
2. Clinically significant abnormal laboratory test values at screening, as determined by the Investigator;
3. Any surgical or medical condition, which in the opinion of the Investigator may pose an undue risk to the subject, interfere with participation in the study, or which may affect the integrity of the study data.
4. Any positive urine drug screen or alcohol test at Screening or clinic admission.
5. Concomitant use of any drugs known to interact with oral absorption or metabolism of pharmaceuticals, including known inducers or inhibitors of cytochrome p450 enzyme system.
6. History of alcohol abuse within 6 months prior to Screening and/or signs or symptoms of alcoholism, as determined by the Investigator.
7. Positive test for Hepatitis B Virus (HBV), Hepatitis C Virus (HCV), or Human Immunodeficiency Virus (HIV);
8. Participation in another clinical trial of an investigational drug (or medical device), or food supplement within 30 days prior to screening, or currently participating in another trial of an investigational drug (or medical device), or food supplement;
9. Donation of greater than 100 mL of either whole blood or plasma within 30 days prior to investigational product administration.
10. Been informed of possible COVID-19 exposure in past 4 weeks, or recent onset of signs or symptoms of possible COVID-19 infection, including cough, shortness of breath, or temperature ≥ 38°C.
11. Traveled via airplane or cruise ship within the last 14 days

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-03-17 (Actual); Primary Completion 2022-05-25 (Actual); Study Completion 2022-05-25 (Actual)

PRIMARY OUTCOMES:
Number, severity, and nature of adverse events following the administration of ascending doses of G3-P01 | Through study completion, up to 70 days
  Evaluating the safety of ascending doses of G3-P01 based on treatment related adverse events
Clinical safety and laboratory parameters- Adverse Events | Through study completion, up to 70 days
  Number of participants with treatment emergent adverse events. Measured by observation and reporting
Clinical safety and laboratory parameters-Clinical Laboratory Results,hematology | Through study completion, up to 70 days
  Number of participants with clinically significant change in clinical laboratory results reported as AEs. Measured by Hematology/Serum Chemistry.
Clinical safety and laboratory parameters-Clinical Laboratory Results, urinalysis | Through study completion, up to 70 days
  Number of participants with clinically significant change in clinical laboratory results reported as AEs. Measured by Urinalysis.
Clinical safety and laboratory parameters-Clinical Laboratory Results, serology | Through study completion, up to 70 days
  Number of participants with clinically significant change in clinical laboratory results reported as AEs. Measured by Serology,
Clinical safety and laboratory parameters-Vital Signs, blood pressure | Through study completion, up to 70 days
  Number of participants with clinically significant change in vital signs reported as AEs. Measured by BP
Clinical safety and laboratory parameters-Vital Signs, pulse | Through study completion, up to 70 days
  Number of participants with clinically significant change in vital signs reported as AEs. Measured by pulse.
Clinical safety and laboratory parameters-Vital Signs, respiratory rate. | Through study completion, up to 70 days
  Number of participants with clinically significant change in vital signs reported as AEs. Measured by respiratory rate.
Clinical safety and laboratory parameters-Vital Signs, body temperature. | Through study completion, up to 70 days
  Number of participants with clinically significant change in vital signs reported as AEs. Measured by body temperature.
Change from baseline in tolerability assessment using Questionnaire | Through study completion, up to 70 days
  Tolerability assessment using the Gastrointestinal Symptom Rating Scale (GSRS). There are 15 individual questions, each with a score of 1-7. Higher scores reflect a worse outcome.
Change from baseline in performance status using Questionnaire | Through study completion, up to 70 days
  Performance status assessment using the Karnofsky Performance Scale Index. The scale is 0-100, with 0 reflecting a worse outcome.

SECONDARY OUTCOMES:
Pharmacokinetic parameters- Cmax | Up to 3 years
  Subject to the development of suitable analytical methods, maximum plasma concentration will be determined.
Pharmacokinetic parameters- Tmax | Up to 3 years
  Subject to the development of suitable analytical methods, time corresponding to the Cmax will be determined.
Pharmacokinetic parameters- AUC | Up to 3 years
  Subject to the development of suitable analytical methods, Area under the plasma concentration-time curve (AUC)" from time zero to the last non-zero concentration (AUC0-t), from time zero till 24-hours post-dose (AUC0-24), from time infinity (extrapolated) (AUC0-inf) will be determined.
Pharmacokinetic parameters- T1/2/ el | Up to 3 years
  Subject to the development of suitable analytical methods, elimination half-life will be determined.
Pharmacokinetic parameters- Vd | Up to 3 years
  Subject to the development of suitable analytical methods, volume distribution will be determined.
Pharmacokinetic parameters- Clr | Up to 3 years
  Subject to the development of suitable analytical methods, renal clearance will be determined.
Pharmacokinetic parameters- dose proportionality | Up to 3 years
  Subject to the development of suitable analytical methods, dose proportionality will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Mazin AlHakim, MD, Principal Investigator — EB FlevoResearch
Locations (1):
- EB FlevoResearch, Almere Stad, Flevoland, Netherlands

IPD SHARING:
Plan to Share IPD: No